CLINICAL TRIAL: NCT01851187
Title: A Randomized Control Study of Prenatal Emotion Management on Maternal Emotion and the Delivery Outcomes
Brief Title: Effect of Perinatal Emotional Management on Maternal Emotion and Delivery Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Y207858
Record Dates: First submitted 2013-05-03; First posted 2013-05-10 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Perinatal Problems; Mental Depression; Complications; Cesarean Section
Keywords: Psychological intervention,; prenatal period,; cesarean section rate,; stage of labor
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- emotional management (EM) group (Experimental): emotional management (EM) group received antenatal psychological intervention
  Interventions: Behavioral: antenatal psychological intervention; Behavioral: routine prenatal care
- the usual care (UC) group (Active Comparator): the usual care (UC) group was given routine prenatal care only
  Interventions: Behavioral: routine prenatal care

INTERVENTIONS:
Behavioral: antenatal psychological intervention — emotion management included:
  (1) Establish relationship between the health care workers and the pregnant women, (2) Determine training objectives, (3) Guide to practice relaxation training, including imagination and abdominal breathing. (4) Make cognitive adjustment, (5) Relieve anxiety and tension by scene simulation and stimulus exposure. (6) Learn emotional self-regulation, (7) Improve self-efficacy by group interaction. (8) Teach prenatal knowledge ,(9) Guide interactive trainings between pregnant women and their couples; (10) Visit delivery rooms.
  Arms: emotional management (EM) group
Behavioral: routine prenatal care — Prenatal routine inspection included blood pressure, weight, uterine fundal height, abdominal circumference, fetal presentation, fetal position, fetal heart rate and so on.

SUMMARY:
Pregnancy or childbirth is a kind of persistent and strong source of stress for pregnant women. Prenatal and intrapartum negative emotions not only damage the mental health of pregnant women, but also have a negative impact on the mode of delivery, labor, postpartum complications and neonatal outcomes . Due to considerations for the effect on the fetus, there is concern of the use of drug treatment for depression during pregnancy. Therefore, psychological interventions have an important role. According to the WHO global survey in Asia 2007-08, China had the highest overall rate of caesarean section (46.2%), and also had the highest rate of caesarean section without indication (11.7%). The embarrassing "first in the world" of caesarean section rate was causing widespread concern in China. Recently, the Chinese government has launched a project named "promoting the rate of natural childbirth and protecting the health of mother and child", trying to reduce the cesarean section rate especially that without medical indication. Therefore, examining if emotional management is effective in reducing negative emotions of pregnant women as well as decreasing the rate of cesarean section is an important research question. Our study aims to help the pregnant women control their anxiety, depressive feelings and other negative emotions by "emotional self-management group training" and we examine if this can reduce the incidence of depression and improve delivery outcomes.

DETAILED DESCRIPTION:
This study tried to explore the effectiveness of prenatal emotional management on pregnant women' delivery outcomes. All participants filled the Questionnaire (PHQ-9) at the baseline assessment. Then they were randomly assigned into the emotional management (EM) group and the usual care (UC) group. The baseline evaluation began at 31 weeks of pregnancy and the mother was followed up to 42 days postpartum. Each subject received the EM package In the EM, and the UC was given only routine prenatal care. PHQ-9 and Edinburgh Postnatal Depression scale（EPDS）were used for assessment.

ELIGIBILITY:
Inclusion Criteria:

1. never have a baby before,
2. with single fetus, head position and normal pelvic measurements,
3. were receiving regular antenatal care,
4. were able to schedule and fulfill questionnaires independently.

Exclusion Criteria:

1. situation with pregnancy complications,
2. surgical history of diseases,
3. current or previous history of any kind of mental disorders.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms assessment | The baseline evaluation began at 31 weeks of pregnancy and the mother was followed up to 42 days postpartum
  All participants were randomly divided into intervention group and control group with 100 in each group. At the baseline assessment, all participants filled the PHQ-9 themselves and instructed by a trained nurse, , the diagnosis of depression was fulfilled by the psychiatrists in our research program. When participants scored over than 10 on the PHQ-9, the diagnostic interview was arranged by a research assistant and was done in one week. At the same time, the results of antenatal physical examination for every participant were collected by our research assistants when a participant was enrolled. After the baseline assessment, participants were randomly assigned into two groups: the emotional management (EM) group and the usual care (UC) group.

SECONDARY OUTCOMES:
Obstetric outcome assessment | after delivery
  Obstetric outcome assessment included the rate of cesarean section, especially the rate without medical indications. The duration of total stage and each stage of labor in natural delivery were concerned.

CONTACTS AND LOCATIONS:
Overall Officials: Hejiang Li, MD, Principal Investigator — The First People's Hospital of Hangzhou
Locations (1):
- The First People's Hospital of Hangzhou, Hangzhou, Zhejiang, China